CLINICAL TRIAL: NCT05200754
Title: A Randomized Open Label Phase-II Clinical Trial With or Without Infusion of Plasma From Subjects After Convalescence of SARS-CoV-2 Infection in High-Risk Patients With Confirmed Severe SARS-CoV-2 Disease
Brief Title: Trial With or Without Infusion of SARS-CoV-2 Antibody Containing Plasma in High-Risk Patients With COVID-19
Acronym: RECOVER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carsten Müller-Tidow (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Institut für Klinische Transfusionsmedizin und Zelltherapie Heidelberg gGmbH (Unknown)
Responsible Party: Sponsor-Investigator, Carsten Müller-Tidow, Medical Director, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SARS-CoV-2CP-HD-001
Record Dates: First submitted 2022-01-20; First posted 2022-01-21 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2 Infection
Keywords: High risk patients; convalescent plasma; post vaccination plasma; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent/Vaccine-boosted Plasma (Experimental): Infusion of plasma on day 1 and 2 (238 - 337 ml anti-SARS-Cov-2 CP/PVP each)
  Interventions: Other: Convalescent/Vaccine-boosted Plasma (CP/PVP)
- Standard of Care (No Intervention): No intervention - standard therapy

INTERVENTIONS:
Other: Convalescent/Vaccine-boosted Plasma (CP/PVP) — Plasma from apheresis obtained from donors, who have recovered from SARS-CoV-2 infection or received a successful vaccination against SARS-CoV-2.
  CP/PVP infusion is administered on two following days. Each CP/PVP bag contains approx. 238 - 337 ml anti-SARS-Cov-2 CP/PVP for infusion.
  Arms: Convalescent/Vaccine-boosted Plasma

SUMMARY:
The study RECOVER is a randomized, open-label, multicenter phase II trial, designed to assess the clinical outcome of SARS-CoV-2 disease in high-risk patients (group 1 to group 4) following treatment with anti-SARS-CoV-2 convalescent/vaccine-boosted plasma or standard of care.

DETAILED DESCRIPTION:
The aim of this randomized phase-II study is to gain evidence on the effect of convalescent plasma/vaccine-boosted plasma in the treatment of SARS-CoV-2 infection in high-risk patients.

High-risk is defined as SARS-CoV-2 positive infection with Oxygen saturation at ≤ 94% at ambient air with additional risk features as categorized in 4 groups:

* group 1, pre-existing or concurrent hematological malignancy and/or active cancer therapy (incl. chemotherapy, radiotherapy, surgery) within the last 24 months or less.
* group 2, chronic immunosuppression not meeting the criteria of group 1
* group 3, age ≥ 50 - 75 years meeting neither the criteria of group 1 nor group 2 and at least one of these criteria: Lymphopenia < 0.8 x G/l and/or D-dimer > 1μg/mL
* group 4, age ≥ 75 years meeting neither the criteria of group 1 nor group 2

The duration of the trial for each patient is expected to be about 3 months, including two days of intervention (infusion of CP/PVP), followed by a follow-up of 3 months. Furthermore viral load is measured in nasopharagyngeal swabs at day 1, 3, 5, 10, 14, 28 or until hospital discharge within 84 days after randomization. Treatment response is assessed daily until day 28, thereafter weekly until day 56, and finally at day 84.

Patients randomized into the standard arm of the study have the possibility to cross over into the experimental arm of the study starting at day 10 (+ 2 days) in case of not improving or worsening clinical condition.

In total 174 patients are planned to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. PCR confirmed SARS-CoV-2 infection in a respiratory tract sample.
2. Oxygen saturation (SaO2) of 94% or less while breathing ambient air or a ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2) of less than 300 mm Hg.
3. High risk due to either pre-existing or concurrent hematological malignancy and/or active cancer therapy (incl. chemotherapy, radiotherapy, surgery) within the last 24 months or less (group 1) and/or chronic immunosuppression not meeting the criteria of group 1 (group 2) and/or Age ≥ 50 -75 years meeting neither the criteria of group 1 nor group 2 (group 3) and at least one of these criteria: Lymphopenia < 0.8 x G/l and/or D-dimer > 1μg/mL and/or Age ≥ 75 years meeting neither the criteria of group 1 nor group 2 (group 4).
4. Blood hemoglobin concentration ≥ 8 g/dl.
5. Provision of written informed consent.
6. Patient is able to understand and comply with the protocol for the duration of the study, including treatment and scheduled visits and examinations.
7. Male or female patient aged ≥ 18 years
8. Postmenopausal or evidence of non-childbearing status. For women of childbearing potential: negative urine or serum pregnancy test within 14 days prior to study treatment.

Exclusion Criteria:

1. Dementia, psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the principle investigator, would affect subject safety and/or compliance.
2. Contraindication to transfusion or history of prior reactions to transfusion blood products.
3. Patients with selective IgA deficiency.
4. Patients with mechanical ventilation and/or extracoporal membrane oxygenation (ECMO) at time of initial inclusion into the trial. Mechanical ventilation is defined as either NIV - non-invasive ventilation or positive pressure ventilation. Enrollment into another clinical trial evaluating specific therapies for COVID-19 is encouraged.
5. Participation in another trial with an investigational medicinal product.
6. Treatment with SARS-CoV-2 convalescent/vaccine-boosted plasma in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | within 84 days
  Time from randomization until an improvement within 84 days defined as two points on a seven point ordinal scale or live discharge from the hospital

SECONDARY OUTCOMES:
Overall survival rate | within 84 days
  Overall survival and overall survival rate at 28, 56 and 84 days
Viral clearance | within 84 days
  SARS-CoV-2 viral clearance and load
Cytokine profiles | within 84 days
  Cytokine changes over time
Antibody titres | within 84 days
  Measurement of antiviral antibody titres
Requirement of mechanical ventilation | within 84 days
  Percentage of patients that required mechanical ventilation
Discharge from hospital | within 84 days
  Time from randomization until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Mueller-Tidow, Prof. Dr., Study Director — University Hospital Heidelberg
Locations (16):
- Germany (16):
  - Charité Universtitätsmedizin Berlin, Berlin
  - Klinikum Bremen-Mitte - Klinik für Innere Medizin I, Bremen
  - Klinikum Chemnitz Medizinische Klinik III, Chemnitz
  - Klinikum Darmstadt Medizinische Klinik II, Darmstadt
  - Universitätsklinikum Dresden Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen Klinik für Infektiologie, Essen
  - Klinikum Frankfurt (Oder) - Medizinische Klinik I, Frankfurt (Oder)
  - Universitätsklinikum Frankfurt Medizinische Klinik II, Frankfurt am Main
  - Universitätsklinikum Freiburg, Allgemeine Infektion-Ambulanz / Klinik für Innere Medizin II, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf Zentrum für Innere Medizin I, Hamburg
  - Universitätsklinikum Heidelberg Innere Medizin V, Heidelberg
  - Thoraxklinik Heidelberg - Studienzentrum Pneumologie, Heidelberg
  - Klinikum Herford, Herford
  - Klinikum Leverkusen - Medizinische Klinik 3, Leverkusen
  - Klinikum Hochsauerland, Meschede
  - Universitätsklinikum Münster Medizinische Klinik B, Münster

IPD SHARING:
Plan to Share IPD: No